CLINICAL TRIAL: NCT06702280
Title: Assessing the Safety of an IGY Supplement on the Gut Microbiome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: IGY Immune Technologies & Life Sciences Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NIMCSF316
Record Dates: First submitted 2024-11-12; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IgY Supplement (Experimental): Participants will ingest the IgY supplement on a daily basis
  Interventions: Dietary Supplement: IgY supplement

INTERVENTIONS:
Dietary Supplement: IgY supplement — Ingesting the immune supplement over the experimental period

SUMMARY:
This study is to evaluate whether Muno-IgY is effective in enhancing immune health among adults over a six week period.

DETAILED DESCRIPTION:
The goal of this single-arm interventional trial is to evaluate the safety and effectiveness of Muno-IGY in a sample population of 20 healthy adults over a six week period. The intervention will be compared to a baseline before ingestion of the supplement with both qualitative questionnaires, a daily diary, and microbiome data gathered by the SIMBA and LIMBA capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old at the inclusion of the study, both female and male subjects.
2. Signed Informed Consent; willing and able to comply with study procedures.
3. Willing to maintain their diet and physical activity levels during the study.
4. Able to swallow a 25mm x 9mm sized capsule

Exclusion Criteria:

1. Use of regular prescription medications, including antihypertensives, anti-inflammatory drugs, corticosteroids, immunosuppressants, antidepressants, antipsychotics, anti-diabetic medications, and anti-arrhythmic agents, which in the opinion of the investigator, would adversely affect study safety or outcome.
2. Prior gastrointestinal disease, surgery, or radiation treatment which, in the Investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion, including, e.g., achalasia, eosinophilic esophagitis, cancer diagnosis or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months before the screening visit is acceptable.
3. History of known structural gastrointestinal abnormalities such as structures or fistulas which may lead to mechanical obstruction.
4. Use of any medications in the week prior to the SIMBA or LIMBA capsule ingestions, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g., opioids, anticholinergics, GLP-1 analogues); laxative and prokinetic use is allowed if it is kept unchanged in the week prior to the SIMBA and LIMBA capsule ingestions. Proton pump inhibitors (PPIs) are allowed provided a wash-out period of 48 hours is respected before swallowing the capsules and PPI treatment is resumed only 4 hours thereafter.
5. Organic motility disorder, including gastroparesis, intestinal pseudo-obstruction, systemic sclerosis, Ogilvie's syndrome.
6. Any significant gastrointestinal, heart, liver, lung, kidney, blood, endocrine or nervous system disease, which in the opinion of the investigator, would adversely affect study safety or outcome.
7. Cancer diagnosis or treatment within the past year (non-melanoma skin cancers are acceptable).
8. History or diagnosis of immunological or infectious disease (hepatitis, tuberculosis, HIV, Parkinson's).
9. History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration.
10. Antibiotic use (except for topical use) ≤ 12 weeks prior to screening. Potential participants may be eligible once a 12-week washout is completed.
11. Consumption of probiotic or prebiotic supplements within 1 month prior to screening. Potential participants may be eligible once a 1-month washout is completed.
12. Any prior Fecal Microbiota Transplantation.
13. Colon cleanses/bowel prep for 2 weeks
14. Pregnant or breastfeeding.
15. Planning to become pregnant.
16. Alcohol or drug abuse.
17. Egg allergy
18. Vegan diet, or other diet where ingestion of eggs is not suitable
19. History of less than 3 bowel movements per week.
20. Are scheduled for an MRI at any time during the study. Potential participants may be eligible to participate once their MRI procedure is completed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | Through study completion (Baseline to the end of the interventional period), an average of 6 weeks
  To assess the safety of Muno-IgY™ in the small intestine. By monitoring the number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Secondary 1 | Through study completion (Baseline to the end of the interventional period), an average of 6 weeks
  Investigate the association or determine if changes in the small and large intestine occur and fecal microbiomes through metagenomic analysis
Secondary 2 | Through study completion (Baseline to the end of the interventional period), an average of 6 weeks
  To assess the bioavailability of the Muno-IgY, using the SIMBA capsule as a tool for sample collection

CONTACTS AND LOCATIONS:
Locations (1):
- Nimble Science, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No